CLINICAL TRIAL: NCT03893331
Title: AcQMap® Global Registry of Procedural and Long-term Clinical Outcomes (AcQMap Registry)
Acronym: DISCOVER
Status: Terminated | Type: Observational
Why Stopped: Sponsor no longer performing clinical studies. Will be only a manufacturing facility
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-AF-006
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Ablation of Arrhythmia's
Keywords: Arrhythmia's

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: AcQMap System — To evaluate procedural and long-term outcomes when using the diagnostic AcQMap System as an imaging and mapping system for ablation of arrhythmias in accordance with the Instructions for Use (IFU).

SUMMARY:
AcQMap Registry is an observational study

DETAILED DESCRIPTION:
AcQMap Registry is an observational, prospective, multi-center, multi-national, open-label registry designed to provide clinical data regarding the commercial, real-life experience with the diagnostic AcQMap System.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Currently scheduled for an ablation of an arrhythmia utilizing the diagnostic AcQMap System.
* Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study.
* Willing and able to give written informed consent.

Exclusion Criteria:

* In the opinion of the Investigator, any known contraindications to an ablation procedure.
* Current enrollment in any study protocol sponsored by Acutus Medical.
* Any other condition that, in the judgment of the investigator, makes the participant a poor candidate for this procedure, the study, or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, extensive travel away from the research center, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any participant 18 years of age or older. Currently scheduled for an ablation of an arrhythmia utilizing the diagnostic AcQMap System.
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Procedural Ablation Outcomes | 12 hours
  • Number of participants who had termination of ablated arrhythmia's to Sinus Rhythm within 12 hours post ablation procedure with or without electrical or pharmacological cardioversion

SECONDARY OUTCOMES:
Long-term Outcome | 3 years
  • First-procedure freedom from any arrhythmia on and/or off AADs, throughout the follow-up period, excluding events in the initial 90 days following the procedure (blanking period).

CONTACTS AND LOCATIONS:
Overall Officials: Simon James, MD, Principal Investigator — James Cook University Hospital
Locations (12):
- I.C.P.S. Hôspital Privé Jacques Cartier, Paris, France
- Klinikum Coburg, Coburg, Germany
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus MC Cardiologie Elektrofysiologie, Rotterdam
- United Kingdom (8):
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Royal Brompton Hospital, London
  - St. George's Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - John Radcliffe Hospital, Oxford
  - Sheffield Teaching Hospital Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided